CLINICAL TRIAL: NCT01109901
Title: Study of Surgical Methods for Cubital Tunnel Syndrome
Brief Title: Comparison of Effect of Anterior Subcutaneous and Submuscular Transposition on Cubital Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213
Record Dates: First submitted 2010-04-19; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2008-10

CONDITIONS: Cubital Tunnel Syndrome
Keywords: Cubital tunnel,subcutaneous transposition,submuscular
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anterior submuscular transposition (Other): it is kind of surgical method
  Interventions: Procedure: Anterior submuscular transposition
- Anterior subcutaneous transposition (Other): it is kind of surgical method
  Interventions: Procedure: anterior subcutaneous transposition

INTERVENTIONS:
Procedure: anterior subcutaneous transposition — transposition of ulnar nerve into subcutaneous bed
  Other Names: ASCT
  Arms: Anterior subcutaneous transposition
Procedure: Anterior submuscular transposition — transposition of ulnar nerve into muscular tissue
  Other Names: ASMT
  Arms: anterior submuscular transposition

SUMMARY:
The purpose of this study is to determine which surgical method is better for cubital tunnel syndrome in outcomes.

DETAILED DESCRIPTION:
Compression of the ulnar nerve at the cubital tunnel is the most common cause of numbness on the ulnar side of the hand. We aimed to compare patient outcomes included pain, sensation, muscle strength and muscle atrophy in two methods of surgery contain Anterior Sub Cutaneous Transposition (ASCT) and Anterior Sub Muscular Transposition (ASMT) of the ulnar nerve in Cubital tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed cubital tunnel syndrome

Exclusion Criteria:

* Significant cervical spine and shoulder disease
* deformity or distortion of the cubital tunnel due to previous trauma to elbow
* recurrent cubital tunnel syndrome after previous surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain | at 6 months post-operatively
  Visual Analogue Scale (VAS) with scores of zero to ten (0 for no pain and 10 intolerable pain) then scored as follows: 0, Sever (8-10); 1, Slight (4-7); 2, none (0-3)

SECONDARY OUTCOMES:
sensation | at 6 months post-operatively
  Sensory disturbance were tested with Semmes-Weinstein filaments and sensory deficits were categorized according to the Yale sensory scale. According to standard scoring system that designed, the severity of sensation and function of the ulnar nerve was scored as follows: 0, Abscent sensation; 1, Decrease or abnormal sensation; 2, Intact sensation.
Muscle strength | at 6 months post-operatively
  Muscle strength was evaluated with the grading system from the Medical Research Council which is based upon a scale of zero to five: 0, No muscle contraction; 1,Flicker or trace of muscle contraction; 2,Limb or joint movement possible only with gravity eliminated; 3,Limb or joint movement against gravity only; 4,Power decreased but limb or joint movement possible against resistance; 5,Normal power against resistance. Then results were scored as follows: 0,Poor (0-1); 1,Moderate (2-3); 2,Good (4-5)
Muscle atrophy | at 6 months post-operatively
  Muscle atrophy was scored with one orthopedic surgeon as follows: 0, sever; 1, moderate; 2, none

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza Shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Iran